CLINICAL TRIAL: NCT01297413
Title: A Phase I/II, Multi-Center, Open-Label Study to Assess the Safety, Tolerability, and Preliminary Efficacy of a Single Intravenous Dose of Allogeneic Mesenchymal Bone Marrow Cells to Subjects With Ischemic Stroke
Brief Title: A Study of Allogeneic Mesenchymal Bone Marrow Cells in Subjects With Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemedica Cell Technologies, Inc. (Industry)
Collaborators: University of California, San Diego (Other); Mercy Gilbert Medical Center at AZ (Unknown); Chandler Regional Medical Center at Chandler AZ (Unknown); UCI Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEM 101-M
Record Dates: First submitted 2011-02-10; First posted 2011-02-16 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Ischemic Stroke
Keywords: allogeneic; adult; stem; cells; stroke; ischemic
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cells (Experimental): All subjects will receive allogeneic adult mesenchymal bone marrow stem cells
  Interventions: Biological: Allogeneic adult mesenchymal bone marrow stem cells

INTERVENTIONS:
Biological: Allogeneic adult mesenchymal bone marrow stem cells — Patients will receive intravenously one dose of 0.5-1.5 million cells per kg of allogeneic adult mesenchymal bone marrow stem cells

SUMMARY:
The purpose of this study is to assess the safety and tolerability of allogeneic adult mesenchymal bone marrow cells administered intravenously to patients with ischemic stroke.

DETAILED DESCRIPTION:
Stroke remains a major global healthcare problem. Recent data compiled by the American Heart Association (AHA) for 2008 show that the annual incidence of new or recurrent stroke in the United States is about 780,000, with approximately 600,000 of these strokes being first attacks. Among adults age 20 and older, the estimated prevalence of stroke in 2005 was 5.8 million in the United States, resulting in >150,000 deaths annually, with 4.8 million stroke survivors alive today. Stroke ranks as the country's third leading cause of death, behind only cancer and heart disease. The only approved treatments of acute ischemic stroke involve restoring blood flow to the affected region by using thrombolytics or mechanical devices that physically remove clots. However, the use of thrombolytics is limited due to the therapeutic window of < 3-6 hours post onset of stroke symptoms such that only a small fraction of stroke patients receive this therapy. Following the completion of a stroke, there is little therapy to offer patients to promote recovery other than physical, occupational, and speech therapy.

Allogeneic mesenchymal stem cells have been used in a number of clinical trials for different indications demonstrated the safety of allogeneic mesenchymal stem cell treatment. In addition to their ability to differentiate into multiple different cell types that would be contributory to the recovery and repair of the brain by replacing destroyed cells, mesenchymal stem cells also secrete angiogenins, cytokines and trophic factors that can support and stimulate multiple other cell types. The cascade of cellular events following the release of these cytokines and trophic factors would also potentially lead to beneficial effects by restoring blood supply, by rescuing cells at risk, and by stimulating the remaining cell populations to repair and propagate new cells and synaptic connections.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke for longer than 6 months
* Brain CT/MRI scan at initial diagnosis and at enrollment consistent with ischemic stroke
* No substantial improvement in neurologic or functional deficits for the 2 months prior to enrollment
* NIHSS score between 6-20
* Life expectancy greater than 12 months
* Prior to treatment patient received standard medical care for the secondary prevention of ischemic stroke
* Adequate organ function as defined by the following criteria:

Exclusion Criteria:

* History of uncontrolled seizure disorder
* History of cancer within the past 5 years.
* History of cerebral neoplasm
* Positive for hepatitis B, C or HIV
* Myocardial infarction withing six months of study entry
* Findings on baseline CT suggestive of subarachnoid or intracerebral hemorrhage within past 12 months.
* Allergies to Bovine or Porcine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-02; Primary Completion 2017-09 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the safety of treatment with aMBMC during the twelve-month study period. | 12 month
  The primary endpoint will be the safety of treatment with aMBMC during the twelve-month study period as determined by the incidence and severity of adverse events, clinically-significant changes on clinical laboratory tests, vital signs, physical and neurologic examinations.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale Score. | 12 months
  The change from the baseline in National Institutes of Health Stroke Scale score will be calculated at 1, 3, 6, 9, 12 months post-treatment, as available:
Mini Mental Status Exam score. | 12 month
  The change from the baseline in Mini Mental Status Exam score will be calculated at 1, 3, 6, 9, 12 months post-treatment, as available.
Barthel Index Score. | 12 month
  The change from the baseline in Barthel Index score at 1, 3, 6, 9, 12 months post-treatment, as available.
The Geriatric Depression Scale Score. | 12 month
  The change from baseline in the Geriatric Depression Scale score at 1, 3, 6, 9, 12 months post-treatment, as available.

CONTACTS AND LOCATIONS:
Overall Officials: Lev Verkh, PhD, Study Director — Stemedica Cell Technologies, Inc.
Locations (3):
- United States (3):
  - Mercy Gilbert and Chandler Medical Center, Gilbert, Arizona
  - University of California Irvine Department of Neurology, Orange, California
  - University of California San Diego Division of Neurological Surgery, San Diego, California

REFERENCES:
- [Derived] Levy ML, Crawford JR, Dib N, Verkh L, Tankovich N, Cramer SC. Phase I/II Study of Safety and Preliminary Efficacy of Intravenous Allogeneic Mesenchymal Stem Cells in Chronic Stroke. Stroke. 2019 Oct;50(10):2835-2841. doi: 10.1161/STROKEAHA.119.026318. Epub 2019 Sep 9. PMID 31495331